CLINICAL TRIAL: NCT01333423
Title: A Phase I With Dose Expansion to Determine the Maximum Tolerated Dose of Liposomal Doxorubicin in Combination With Seliciclib for the Treatment of Patients With Metastatic Triple Negative Breast Cancer
Brief Title: Maximum Tolerated Dose (MTD) of Liposomal Doxorubicin in Combination With Seliciclib for Patients With Metastatic Triple Negative Breast Cancer (TNBC)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0013; 1R01CA152228-01A1 (NIH)
Record Dates: First submitted 2011-04-08; First posted 2011-04-12 (Estimated); Last update posted 2012-06-26 (Estimated); Status verified 2012-06

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Metastatic Triple Negative; ER/PR/HER2 negative; Locally advanced; Stage IV; Metastatic; Seliciclib; Liposomal Doxorubicin; Doxil; Doxorubicin Hydrochloride (Liposomal)
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms; Neoplasm Metastasis | interventions — liposomal doxorubicin; Doxorubicin; Liposomes; Roscovitine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Doxil + Seliciclib (Experimental): Doxil (Liposomal doxorubicin) 40 mg/m2 intravenous (IV) over 2 -3 hours on Day 4 and Seliciclib starting dose 200 mg orally twice a day on Days 1 - 3 of 28 day cycle
  Interventions: Drug: Liposomal Doxorubicin; Drug: Seliciclib

INTERVENTIONS:
Drug: Liposomal Doxorubicin — 40 mg by vein administered over 2 -3 hours on Day 4 of a 28 day cycle.
  Other Names: Doxil; Doxorubicin Hydrochloride (Liposomal)
Drug: Seliciclib — Starting dose 200 mg by mouth twice daily on Days 1 - 3 of a 28 day cycle.

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of seliciclib that can be given in combination with liposomal doxorubicin to patients with metastatic breast cancer.

DETAILED DESCRIPTION:
The Study Drugs:

Seliciclib is designed to stop cancer cells from dividing, which may cause them to die.

Doxorubicin is a chemotherapy drug that is designed to stop the growth of cancer cells, which may cause the cells to die. Liposomal doxorubicin is a redesigned version of doxorubicin. The drug, doxorubicin, is enclosed in a fat bubble called a liposome. This is designed to allow the drug to get into the tumor tissue better and to stay in the body for a longer time.

Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a dose level of seliciclib based on when you joined this study. Up to 6 dose levels of seliciclib will be tested. At least 2 participants will be enrolled at each dose level. The first group of participants will receive the lowest dose level. Each new group will receive a higher dose than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of seliciclib is found.

All participants will receive the same dose level of liposomal doxorubicin.

Drug Administration:

You will take seliciclib by mouth with a cup (8 ounces) of water twice a day on Days 1-3 of each 28-day study cycle. The 2 doses should be taken 12 hours apart. Seliciclib should be taken 1 hour before or 2 hours after a meal. If you miss a dose, it can be taken up to 2 hours after the scheduled time. If it has been more than 2 hours, the missed dose should not be taken. You should resume taking the study drug at the next normally scheduled time.

You will receive liposomal doxorubicin by vein over 2-3 hours on Day 4 of each cycle.

On Days 5-28 you will not receive any study drugs.

Study Visits:

At all study visits, you will be asked about any side effects you may be having and about any other drugs you may be taking.

On Day 1 of every cycle:

* You will have a physical exam, including measurement of your weight and vital signs.
* Your performance status will be recorded.
* Blood (about 1-2 teaspoons) and urine will be collected for routine tests.

During Week 2 of Cycle 1:

-Blood (about 1-2 teaspoons) will be drawn for routine tests.

You will have an ECHO or MUGA scan at least every 4 cycles to check your heart function.

After every even-numbered cycles (Cycles 2, 4, 6 and so on), you will have either a CT or MRI scan to check the status of the disease.

Length of Study:

You may continue taking the study drugs for as long as the doctor thinks it is in your best interest. You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over once you have completed the end-of-study visit.

End-of-Study Visit:

About 4-6 weeks after you have stopped receiving the study drugs, you will have an end-of-study visit. The following tests and procedures will be performed:

* You will have a physical exam, including measurement of your weight and vital signs.
* Your performance status will be recorded.
* Blood (about 1-2 teaspoons) and urine will be collected for routine tests.
* You will be asked about any symptoms you may be having and drugs you may be taking.

This is an investigational study. Seliciclib is not FDA-approved or commercially available. It is currently being used for research purposes only.

Liposomal doxorubicin is FDA-approved and commercially available for metastatic breast cancer. The use of these drugs together is investigational.

Up to 40 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Both male and female patients with invasive cancer that is confirmed ER/PR/HER2 negative carcinoma of the breast with locally advanced or stage IV disease that is not amenable to curative therapy. For purposes of this study, triple negative disease will be tumors that have ER/PR <10% and HER2 </=1+ by IHC or HER2 FISH non-amplified (ratio <2.0).
2. Patients must have an ECOG performance status of 0, 1 or 2
3. Age >/= 18 years
4. Women must not be pregnant or lactating because of the teratogenic potential of these drugs. All females of childbearing potential (i.e. A female not free from menses > 1 year or not surgically sterilized) must have a blood test or urine study within 2 weeks prior to start of therapy to rule out pregnancy.
5. Women of childbearing potential (i.e. A female not free from menses > 1 year or not surgically sterilized) and are strongly advised to use an accepted and effective non-hormonal method of contraception.
6. Must have at least one site of objective measurable or evaluable disease. Baseline measurements and evaluations must be obtained within 4 weeks of start of therapy.
7. Patients must be disease free of prior malignancy for >/= 5 years with the exception of curatively treated squamous cell carcinomas of the skin or carcinoma in situ of the cervix or breast.
8. Patients must have no serious medical illness, other that treated by this study, which would limit survival to less than 1 month or psychiatric illness which would limit informed consent.
9. Patients must not have peripheral neuropathy > grade 2.
10. Required Cardiac Parameters: Patients must not have had a history of New York Heart Association class 3 or 4 heart failure, or history of myocardial infarction, unstable angina or CVA within 6 months of protocol registration. LVEF > 50% by MUGA or ECHO.
11. Patients must not have history of PR prolongation or AV block
12. Required laboratory parameters: Patients must have serum creatinine < 1.5 mg/dl.
13. Patients must have adequate hematologic functions: granulocytes > 1500/mm^3 and platelets > 100,000/mm^3
14. Patients must have adequate hepatocellular function: SGOT (AST) and SGPT (ALT) < 1.5 x upper limit of normal (unless liver is involved by tumor, in which case SGOT (AST) and SGPT (ALT) can be < 2.0 x upper limit of normal)
15. Patients must have no history of prior therapy with seliciclib.
16. Patients must not have received a cumulative dose of doxorubicin of greater than 360 mg/m^2 or epirubicin of greater than 640 mg/m^2. Patients who have received >240 mg/m^2 of doxorubicin or >400 mg/m^2 of epirubicin should be advised to undergo evaluation of left ventricular ejection fraction (LVEF) with echocardiogram (ECHO) or gated heart scan (MUGA) prior to initiating therapy.
17. Concurrent use of hormonal therapy is not permitted. Concurrent radiation therapy is not permitted.
18. Patients must not have had prior organ allograft or require immunosuppressive therapy.
19. Patients must have completed and recovered from the effects of prior chemotherapy (</= grade 2 toxicity).
20. Patients must have received at least one prior chemotherapy regimen for metastatic disease. Progression within 6 months of adjuvant chemotherapy will be considered equivalent to one prior chemotherapy for metastatic disease.

Exclusion Criteria:

1) None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-09; Primary Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with a Dose Limiting Toxicity(DLT) | Cycle 1 of therapy (28 days)
  Dose-limiting toxicity (DLT) defined as NCI Common Toxicity Criteria (version 4.0): Grade 3 or 4 thrombocytopenia lasting > 2 weeks; Grade 3 or 4 neutropenia lasting >2 weeks; Febrile neutropenia; Grade 3 or 4 non-hematologic toxicity that lasts > 72 hours despite appropriate medical management (excluding grade 3 fatigue); or Delay in administration of cycle 2 of therapy for >2 weeks due to myelosuppression. DLT must be considered treatment related and occur during cycle 1 of therapy.

SECONDARY OUTCOMES:
Number of Participants with Clinical Response | 6 months
  Disease response assessed using standard imaging techniques every two cycles. Response measured and defined using modified RECIST criterias of CR, PR or SD at 6 months where Complete Response (CR): Disappearance of all target lesions; Partial Response (PR): At least a 30% decrease in sum of longest diameter of target lesions, taking as reference baseline sum longest diameter; and Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for Progressive Disease (PD), taking as reference smallest sum of longest diameter since treatment started.

CONTACTS AND LOCATIONS:
Overall Officials: Stacy Moulder, MD, Principal Investigator — UT MD Anderson Cancer Center

REFERENCES:
- See also: UT MD Anderson Website — http://www.utmdanderson.org